CLINICAL TRIAL: NCT06482411
Title: Exploration of Effect Weight Loss Outcome Related to Factors After Treatment of Weight Loss (WRRFA).
Brief Title: Risk Factors Affect Weight Loss Outcomes After Treatment.
Acronym: WRRFA
Status: Completed | Type: Observational
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Chen,Chung-Yen, Deputy Administrative Offices Director, E-DA Hospital
Other Study IDs: EMRP19113N
Record Dates: First submitted 2024-06-17; First posted 2024-07-01 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Weight Regain
Keywords: Obesity; Weight regain; Bariatric surgery; Anti-obesity medications; Lifestyle intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-Surgical group: Participants were treated with anti-obesity medications plus lifestyle intervention therapy Participants were treated with TFDA-approved anti-obesity medications (e.g. Saxenda, Contrave, etc.).
- LSG: Bariatric surgery group(Restriction procedure): Laparoscopic Sleeve Gastrectomy
- OAGB: Bariatric surgery group(Restriction procedure): One anastomosis gastric bypass
- SASI: Bariatric surgery group(Restriction procedure): Single Anastomosis Sleeve Ileal Bypass

SUMMARY:
The treatment for weight loss was more diverse due to the higher prevalence of obesity. In addition to weight loss medications, many patients seek bariatric surgery to treat obesity. Although bariatric surgery was the most effective way, the patients still get weight gain due to failure to control their lives. The failure weight loss is caused by complex risk factors, such as dietary habits, quality of life, physical inactivity, comorbidities remission rate, and more related to the failure weight loss factors. To explore weight gain factors, the study uses many questionnaires, including demographic parameter and exercise frequency survey, the WHOQOL-BREF assessment, The Bariatric Quality of Life Questionnaire (BQL), the Three-Factor Eating Questionnaire (TFEQ-R18), the Yale Food Addiction Scale version 2.0 (YFAS 2.0), and Depression Anxiety Stress Scales-21 (DASS-21). The investigators assess different factors like quality of life, food addiction, preferences, psychological status, and regular examination parameters to identify reasons for unsuccessful weight loss. The study aims to establish the model for the prediction of risk factors after treatment of weight loss so that the tools will help to manage the best weight control for the future.

DETAILED DESCRIPTION:
Obesity is a disease worldwide. Hence, many patients seek many different treatments for obesity. The methods for obesity include medical and surgical treatment. The medicine treatment indication for diabetes previously increased indication to weight loss for obese patients now. Recently, the four approved weight loss medicines by the Taiwan Food and Drug Administration (TFDA) include Orlistat, Liraglutide, Contrave, and Semaglutide. In addition to medications for weight loss, indications for more than 30 body mass index (BMI) and more than 27 BMI with uncontrol obesity-related comorbidities.

Another weight loss treatment was bariatric surgery. The surgical treatment focuses on morbidity obese patients. Decrease food intake and absorb calories by changing the structure of the stomach and intestine to weight loss and improve comorbidities. Moreover, three functions for bariatric surgery by different mechanisms to weight loss outcome, include (1) restriction, (2) malabsorption, (3) mixed function, and which indication for more than 37.5 BMI and more than 32.5 BMI with two or more uncontrol obesity-related comorbidities.

Since obesity is not a condition that can be cured by surgical removal of lesions forever, patients often experience weight loss failure after receiving both medical and surgical treatments. Particularly, the probability of weight loss failure after medical treatment is higher than that after surgical treatment. Complexed risk factors caused failure weight loss from behavioral dietary, quality of life, remission rate of comorbidities, genetic inheritance, physical Inactivity, and psychological status. Moreover, failure weight loss has two definitions (1) weight regain (WR) and (2) insufficient weight loss (IWL). The investigators searched many studies to organize failure weight loss definitions referenced by Surgery for Obesity and Related Disease (SORD) in the American Society for Metabolic and Bariatric Surgery (ASMBS). IWL is defined as less than 50 percent excess weight loss (%EWL) or less than 35 BMI after 18 months. WR is defined as (1) more than the nadir weight of 10 kg (2) more than the nadir weight of 25% EWL (3) more than the nadir weight of 5 BMI (4) successfully reduced to a BMI below 35, but after 1-year post-treatment, it exceeded BMI 35 (5) at any point within 1-year post-treatment, the weight is higher than the lowest weight achieved. (6) the weight regained is more than 15% of the lowest weight achieved. In contrast to weight gain after medicine which is defined by population proportion 5%, 10%, 15%, 20% statistical analysis.

The study was an observational cohort study. The investigators will use the six types of questionnaires (1) Demographic parameters and exercise frequency (2) WHOQOL-BREF scale (3) Bariatric Quality of Life Questionnaire (BQL) (4) Three-Factor Eating Questionnaire (TFEQ-R18) (5) Yale Food Addiction Scale (YFAS)2.0 (6) Depression Anxiety Stress Scales-21 (DASS-21). Approximately 5,000 adults who underwent bariatric surgery between January 2017 and December 2024 have been identified for inclusion. The investigators hypothesize that these risk factors are significantly interrelated and are associated with suboptimal weight loss or weight regain following surgery. The primary aim is to analyze the risk of weight regain across different bariatric treatments and identify factors that can support long-term, quality weight management.

ELIGIBILITY:
Inclusion 1.65 ≥ Age ≥ 20 years-old. 2.BMI ≥ 30. 3.Once attempted exercise or dietary control. 4.No cognitive deficiency and clear communication. 5. No severe psychotic disorders were evaluated by the psychiatrist. (e.g. schizophrenia, bipolar disorder, or severe depression).

6. Signing the informed consent form for clinical trials.

Exclusion

1. Once underwent bariatric surgery.
2. Once used the GLP-1 receptor agonist.
3. Pregnancy or preparation for pregnancy.
4. Once and presenting gastric cancer.
5. Presenting the other cancer.
6. The abnormal endocrine system causes diseases with obesity.
7. Major organ abnormalities (e.g., kidney failure, liver failure, heart failure, etc.).
8. Gastric ulcer, and severe gastroesophageal reflux.
9. Severe psychiatric disorders (schizophrenia, severe bipolar disorder, and depression, etc.).
10. Bulimia nervosa or anorexia nervosa.
11. Drug and alcohol abuse.
12. Helicobacter pylori is not for bariatric surgery.
13. The following diseases or conditions preclude the use of Contrave: 1)Uncontrolled hypertension, 2) History or current diagnosis of epilepsy, 3) Allergy to this medication, 4) Medications evaluated by a physician to interact with this drug (antidepressants, antipsychotics, liver medications, heart medications).
14. The following diseases or conditions preclude the use of GLP-1 medication: 1) History or current diagnosis of medullary thyroid carcinoma, 2)History or current diagnosis of Multiple Endocrine Neoplasia syndrome type 2, 3)Allergy to this medication, 4)Medications evaluated by a physician to interact with this drug (antidepressants, antipsychotics, liver medications, heart medications).
15. The following diseases or conditions preclude the use of Xenical medication: 1) History or current diagnosis of cholestasis, 2) Allergy to this medication, 3) Medications evaluated by a physician to interact with this drug (antidepressants, antipsychotics, liver medications, heart medications).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: More than 30 BMI obese patients consent to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 3602 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
The proportion of failure weight loss | Month 6, Year 1, Year 1.5, Year 2
  Compare the proportion of failure weight loss after bariatric surgery and medication plus life intervention at 1, 1.5, and 2 years.

SECONDARY OUTCOMES:
The percentage of total weight loss changes | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in percentage of total weight loss
Weight change | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in weight change
BMI change | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from BMI in weight change
Exercise change | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from baseline in exercise frequency
Physiological parameter change | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from baseline in physiological parameter.
  1. Concentration of blood sugar test, such as fasting blood glucose (mg/dL), HbA1c (%), C-peptide (ng/dL), Insulin (μIU/mL).
  2. Concentration of blood lipid test, such as total choleserol (mg/dL), TG (mg/dL), HDL-C (mg/dL), LDL-C (mg/dL). Concentration of liver and renal function test, such as ALT (U/L), AST (U/L), eGFR (mL/min/1.73m2), creatnine (mg/dL).
  3. Concentration of urine and anemia test, such as uric acid (mg/dL), hemoglobin (g/dL), HCT (%), Fe (ug/dL).
  4. Concentration of micro-nutrient test, such as IPTH (pg/mL), Ca (mEq/L), Zinc (ug/dL).
  Above all, the biochemistry with patients at the hospital.
The comorbidity remission rate. | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from baseline in proportion of comorbidity remission
Complication events. | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from baseline in proportion of Complication events
Health quality of life change | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in World Health Organization Quality-of-Life Scale (WHOQOL-BREF).The questionnaire has 28-items and belong to four domains (physical, psychological, social, quality of life). Use a Likert-type five-point scale, and higher the score, the better the quality of life. The 4 domain scores are each converted into a scale from 0 to 100.
Quality of life after weight loss treatment change | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in Bariatric Quality of Life Questionnaire (BQL). The questionnaire consists of two main parts and has 15-items. Obesity comorbidities and complications after treatment.The factors related to quality of life. The total score of both parts ranges from 0 to 78, with a higher score indicating better quality of life.
Eating behavior | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in Three-Factor Eating Questionnaire (TFEQ-R18). The questionnaire has 18-items and consist three domains (1) Cognitive Restraint (CR), (2) Uncontrolled Eating (UE), and (3) Emotional Eating (EE). Use a Likert-type four-point scale, and the total score ranges from 18 to 72, with the higher score, prefer the domain.
Food addiction | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in Yale Food Addiction Scale (YFAS)2.0. The questionnaire has 25-items. Absence of food addiction: 0-1 point. Mild food addiction: 2-3 points. Moderate food addiction: 4-5 points. Severe food addiction: ≥ 6 points. Higher score indicating poorer control to food eat.
Psychiatric status | Follow-up 8 times (Baseline, Month 1, Month 3, Month 6, Month 9, Year 1, Year 1.5, Year 2) visit for all secondary outcome
  Change from Baseline in Depression Anxiety Stress Scales-21 (DASS-21). The questionnaire has 21-items and consist three domains. Depression domain has score rang of 0-14 points. Higher score has severe depression. Anxiety domain has score rang of 0-10 points. Higher score has severe Anxiety. Stress domain has score rang of 0-17 points. Higher score has severe Stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Yen Chen, Kaohsiung City, Yanchao District, Taiwan